CLINICAL TRIAL: NCT05869929
Title: Health Effects of Supplementation With Vegetables
Brief Title: Easy Peasy: Health Effects of Supplementation With Vegetables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ann Skulas-Ray, Assistant Professor of Nutritional Sciences, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Easy Peasy
Record Dates: First submitted 2023-02-23; First posted 2023-05-22 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior | interventions — Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegetables (Experimental): 4-5 servings of vegetables daily, per USDA definition.
  Interventions: Dietary Supplement: Vegetables
- Normal diet (No Intervention): Participant maintains normal diet, no intervention

INTERVENTIONS:
Dietary Supplement: Vegetables — 4-5 servings of vegetables daily, per USDA guidelines.
  Arms: Vegetables

SUMMARY:
The proposed study aims to test the effects of supplementing healthy individuals (with low baseline vegetable consumption) with 5 servings of vegetables (80-120g per serving) per day for 4 weeks on blood lipids and other cardiometabolic outcomes. Previous studies indicate the potential to see significant effects in this population and within this amount of time. Importantly, the investigators will also be including a weekly cooking demonstration as part of the intervention, which provides an essential hands-on participatory component and allows participants to connect with one another in a group setting, which aids in acceptability and adherence to dietary interventions. The investigators hypothesize that 4 weeks of daily supplementation with 4-5 servings of vegetables will significantly improve LDL-C and other cardiometabolic outcomes in healthy adults.

ELIGIBILITY:
Inclusion criteria:

* 18-65 years of age
* Consuming a typical American diet (i.e. not engaged in a structured diet)
* Willing and able to eat vegetables provided (i.e. not allergic or adverse to vegetables provided).

Exclusion criteria:

* Pregnant or lactating
* Participants who currently eat 5+ servings/cups of vegetables per day (excluding tomato paste/sauce, and fried potatoes 'French fries')
* Any condition that would interfere with the participant's data, at the study team's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
LDL-C/non-HDL-C | 4-6 weeks
Brachial and central blood pressure | 4-6 weeks
  systolic and diastolic pressures

SECONDARY OUTCOMES:
Augmentation Index | 4-6 weeks
  augmentation index corrected for heart rate augmentation index corrected for heart rate
Other lipids and lipoproteins | 4-6 weeks
  HDL-C, total cholesterol, and triglycerides
Glucose | 4-6 weeks
  Fasting blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Ann Skulas-Ray, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No